CLINICAL TRIAL: NCT05034679
Title: Wether Corona Vaccination Has Negative Impact on AMH- Anti Mullerian Hormone Which Express Ovarin Function
Brief Title: Impact of Corona Vaccination on AMH- Anti Mullerian Hormone
Acronym: Israel
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Eran Horowitz M.D., Senior Physician, Wolfson Medical Center
Other Study IDs: 0013-21-WOMC
Record Dates: First submitted 2021-08-29; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Patient Participation
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples evaluated for Anti Mullarin Hormone (AMH)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vaciinated: First group patients who vaccinated and measure the AMH before and up to 9 months after vaccination.
  Interventions: Biological: Vcinated
- Infected patients by covid-19 and not vacinated: Second group patients who were infected by Covid-19 ant therefor were not vaccinated
- Not infected nor vacinated: Ptients who who were not infected nor vacinated by Covid-19.

INTERVENTIONS:
Biological: Vcinated — Patients who were vacinated.
  Groups: Vaciinated

SUMMARY:
Since December 2020 Nationwide anti-COVID-19 vaccination began in Israel using the Pfizer - BioNtech vaccine (BNT162b2 mRNA). The vaccination campaign has been associated with concerns regarding potential detrimental effects on future fertility. The aim of the study is to determine the impact of COVID-19 vaccination on n AMH- Anti Mullerian Hormone which express ovarin function.

disease and/or immunization on human follicular function, by comparing follicular steroidogenesis, response to the LH/hCG trigger, and oocyte quality biomarker (HSPG2), in the aspirated follicular fluid of patients undergoing ovum pick-up.

DETAILED DESCRIPTION:
Our assumption is that there is no effect of the vaccination on the AMH level. We plan to recruit 90 patients who are divided to three groups First group patients who vaccinated and measure the AMH before and up to 9 months after vaccination. Second group patients who were infected by Covid-19 ant therefor were not vaccinated to compare the AMH level before and after the infectious. The third group patients who were not infected and not vaccinated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-44

Exclusion Criteria:

Age over 45

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women in reproductive age.
Study Population: Women who are going through IVF treatments.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
Amh levels | 9 months
  Before and after vacination

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson medical center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No